CLINICAL TRIAL: NCT02435394
Title: Web System for Engaging Families & Doctors in Continuous Asthma Quality Improvement
Acronym: Asthma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: After IRB review, this study is no longer considered a clinical trial
Sponsor: Total Child Health, Inc. (Industry)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R44HL117482 (NIH)
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Remote Coach plus Asthma Module (Experimental): The intervention is for practices to have remote coach support for patients with asthma in addition to doctors using CHADIS-Asthma module. Practices will start sequentially for a time series analysis.
  Interventions: Behavioral: Remote Coach plus Asthma Module
- Asthma Module- No Coach (Experimental): The intervention is for practices to use CHADIS-Asthma module to improve patient care without a remote coach assisting patient adherence.
  Interventions: Behavioral: Asthma Module- No Coach
- CHADIS- no Asthma module (Active Comparator): Practices using CHADIS but no Asthma module as a control condition.
  Interventions: Behavioral: CHADIS- no Asthma Module

INTERVENTIONS:
Behavioral: Remote Coach plus Asthma Module — The intervention is for a remote coach to assist patients with asthma for practices which will use Asthma module for guidance for asthma care.
  Other Names: Remote Coach
  Arms: Remote Coach plus Asthma Module
Behavioral: Asthma Module- No Coach — The intervention is for practices to use the Asthma module for guidance for asthma care without assistance by a remote coach.
  Arms: Asthma Module- No Coach
Behavioral: CHADIS- no Asthma Module — The practices will use the general CHADIS tool without access to the Asthma Module add-on to assist in asthma care.
  Arms: CHADIS- no Asthma module

SUMMARY:
Asthma, one of the most common pediatric illnesses, is optimally managed according to National Heart Lung and Blood Institute (NHLBI) guidelines yet this is not often done in primary care. This project is to develop and test the effects of using a module for guideline based care in the Child Health and Development Interactive System (CHADIS) online system by prompting and incorporating patient symptom/control and adherence data from standard questionnaires to inform visits and providing automated patient specific education and Asthma Action Plans in individual Care Portals.

DETAILED DESCRIPTION:
We will complete the formative work collecting professional opinion to create and pilot the initial CHADIS Asthma Intervention module (CHADIS-AI), an innovative decision support system. CHADIS-AI content will be assembled and vetted by asthma experts and primary care providers (PCPs). Parent and teen focus groups will vet the content and language of the adherence materials and Care Portal. A system will also be established for points for patient participation, to give clinicians Maintenance of Certification (MOC) credit, and ongoing run chart reports of their patients' asthma status for continual Quality Improvement (QI) feedback. The resulting system will be pilot tested and refined by clinician feedback. Practices will be randomly assigned to intervention vs control. Control practices will use CHADIS for asthma care without the A-I module. Intervention practices will be further randomized to have remote coach support for patients or not. Outcomes will be examined of asthma severity/control, match of severity with guideline based medication management, numbers of Emergency Department (ED) visits, hospitalizations and oral steroid use. Effect of remote coaching will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis

Exclusion Criteria:

* Not English or Spanish speaking

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
NHLBI recommended controller meds used | 3-12 months
  match between severity rating and NHLBI recommended med mgt

SECONDARY OUTCOMES:
Emergency department visits | 3-12 months
  Self reported interval ED visits
Asthma trigger mitigation | 3-12 months
  self-reported efforts to reduce asthma triggers
Hospitalizations for asthma | 3-12 months
  Self reported hospitalizations
Steroid bursts | 3-12 months
  Self reported use of steroid bursts for asthma exacerbations
Influenza vaccine receipt | 3-12 months
  self reported receipt of flu vaccine for this season
asthma symptom control | 3-12 months
  severity/control ratings

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Howard, MD, Principal Investigator — Total Child Health
Locations (1):
- Total Child Health, Baltimore, Maryland, United States